CLINICAL TRIAL: NCT00204295
Title: Phase 2 Study on Brain Tumor Uptake of the Amino Acid O-(2-[F-18]Fluorethyl)-L-Tyrosin (FET)
Brief Title: Study on Amino Acid Uptake in Brain Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FET-HT-MS
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Brain Neoplasms
Keywords: Brain neoplasms; Positron-Emission Tomography; Amino Acids; Magnetic Resonance Imaging
MeSH Terms: conditions — Brain Neoplasms | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

INTERVENTIONS:
Drug: O-(2-[F-18]Fluorethyl)-L-Tyrosin (FET) - PET

SUMMARY:
The purpose of this study is to determine the uptake of the amino acid O-(2-[F-18]Fluorethyl)-L-tyrosin (FET) in human brain tumors using positron emission tomography. A comparison to MRI and histopathological samples is used.

DETAILED DESCRIPTION:
Radioactively labelled amino acids have been used for years to delineate primary brain tumors and for the early detection of tumor recurrence. Positron emission tomography studies indicate that the extent of amino acid uptake correlates to the true histological extent of gliomas. Recently a fluorine-18 labelled amino acid has been introduced (O-(2-[F-18]Fluorethyl)-L-tyrosin (FET)), which is suitable for routine use in brain tumor patients. There is evidence that this amino acid is transported into brain and brain tumors by the amino acid transport of the L-type. The cDNA of this L-transporter has recently been cloned and has been shown to be identical to the light chain of the 4F2-antigen (CD98), which has previously been described as marker of cell growth and proliferation.

The heavy chain of this heterodimer is known to modulate integrins which are thought to play a fundamental role in glioma invasion.

Besides the evaluation of the diagnostic capability of FET in brain tumors, a comparison of FET uptake in vivo and CD98 expression ex-vivo is performed with tissue slices as available after routine surgery in glioma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected primary brain tumors
* CT or MRI showing lesion of >= 2,5 cm
* Any age; parents informed consent in children available
* Karnofsky-Index >= 20 %
* Referral by Depts. of Neurology, Neuro-Oncology, Neurosurgery, or Pediatric Neurology at the UKM
* Biopsy and/or surgery planned
* Patient is able to lie during the PET scan for 50 minutes without moving • Patient must be able to give informed consent; signature must be present before the PET scan

Exclusion Criteria:

* Pregnancy or breast feeing
* Patients, who by psychiatric disease are not able to give informed consent
* Complete renal failure
* Inclusion to other studies according to § 23 of the German radiation protection law

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2004-01

PRIMARY OUTCOMES:
Histological samples where available
CD98 staining where available

SECONDARY OUTCOMES:
Clinical follow-up for at least one year

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Weckesser, MD, Principal Investigator — Department of Nuclear Medicine, University Hospital Muenster
Locations (1):
- Department of Nuclear Medicine, University Hospital Muenster, Münster, North Rhine-Westphalia, Germany